CLINICAL TRIAL: NCT06658561
Title: Efficacy and Safety Research of Cold Snare Polypectomy and Hot Snare Polypectomy in the Treatment of 4-9 mm Diameter Colorectal 0-Isp and 0-Ip Polyps: a Prospective, Multicenter, Randomized Controlled Study(FAST -REST Study)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Jinshan Hospital Fudan University (Other); Second Affiliated Hospital of Soochow University (Other); The Third People's Hospital Yunnan (Unknown); People's Hospital Mojiang (Unknown); Shanghai Yueyang Integrated Medicine Hospital (Other); Huadong Hospital (Other)
Responsible Party: Principal Investigator, ZOU DUOWU, Director of Gastroenterology Department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RuijinH20241532
Record Dates: First submitted 2024-07-18; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Cold Snare Resection; Hot Snare Resection; Polyps of Colon
Keywords: cold snare resection; hot snare resection; colorectal Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold snare polypectomy group (Other): 1. Rotate the lens body to make the polyp at about 6 o'clock.
  2. Place the special cold snare in the normal mucosa 1-2mm away from the polyp edge.
  3. Tighten the snare at a constant speed and gently lift it up.
  4. Excision.
  5. According to the polyp size, use the colonoscope suction channel or directly use the snare to pull out the tissue for further pathological examination.
  6. Piecemeal resection will be performed if the en-bloc resection fails.
  Interventions: Procedure: cold snare polypectomy
- hot snare polypectomy group (Other): 1. Rotate the lens body to make the polyp at about 6 o'clock.
  2. According to evaluation of the polyps, directly place the snare on the edge of the polyp including a clear margin of normal tissue (1-2 mm) or after submucosal injection.
  3. Tighten the snare at a constant speed and gently lift it up.
  4. Use the electrocoagulation and electroscission mode, power on for several seconds until the polyp is cut off.
  5. According to the polyp size, use the colonoscope suction channel or directly use the snare to pull out the tissue for further pathological examination.
  6. Piecemeal resection will be performed if the en-bloc resection fails.
  Interventions: Procedure: hot snare polypectomy

INTERVENTIONS:
Procedure: cold snare polypectomy — Place the special cold snare in the normal mucosa 1-2mm away from the polyp edge. Tighten the snare at a constant speed and gently lift it up and then excision.
  Other Names: CSP
  Arms: cold snare polypectomy group
Procedure: hot snare polypectomy — According to evaluation of the polyps, directly place the snare on the edge of the polyp including a clear margin of normal tissue (1-2 mm) or after submucosal injection. Tighten the snare at a constant speed and gently lift it up.Use the electrocoagulation and electroscission mode, power on for several seconds until the polyp is cut off.
  Other Names: HSP
  Arms: hot snare polypectomy group

SUMMARY:
This study will evaluate the efficacy and safety of cold snare polypectomy(CSP) and hot snare polypectomy(HSP) in the treatment of colorectal 4-9mm 0-Isp and 0-Ip polyps, and compare the complete resection rate, postoperative late bleeding rate, intraoperative bleeding rate, en bloc resection rate, operation time and the number of metal clips used. The conclusion of this study will help clinical doctor develop more effective resection strategies for colorectal 0-Isp and 0-Ip polyps, and provide more effective treatment for patients.

DETAILED DESCRIPTION:
Colorectal polyps are one of the precancerous lesions of colorectal cancer, 60-80% of which eventually become advanced colorectal cancer. Therefore, early resection of colorectal polyps can effectively reduce the incidence of colorectal cancer. Polyps under white light are judged mainly according to the shape, size and color of polyps. At present, the Paris classification is often used to divide 0-I uplifted polyps into sessile polyps (0-Is), sessile-pedunculated polyps (0-Isp) and pedunculated polyps (0-Ip). It is generally believed that there are thick arteries in 0-Ip polyps, especially thick pedunculated polyps, which are prone to uncontrollable bleeding during operation. 0-Is polyps have small scattered blood vessels and low intraoperative bleeding risk, while the morphological and structural characteristics of 0-Isp polyps are between the two. The current guidelines recommend HSP for 0-Isp and 0-Ip polyps <1 cm, but the internal blood vessels of these polyps are not thick. There is no guidance on whether they can be resected by CSP method, and there is a lack of prospective large sample clinical research. This study will include0-Isp /0-Ip polyps <1cm, and observe the safety and effectiveness of CSP for the above polyp resection , so as to provide reference for the clinical treatment of colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old, male or female
2. At least one polyp with size of 4-9 mm 0-Isp or 0-Ip is found during colonoscopy
3. Voluntarily sign informed consent for endoscopic treatment

Exclusion Criteria:

1. Boston Bowel Preparation Scale<6 points.
2. Patients who receive antiplatelet/anticoagulant therapy within 5 days before polypectomy.
3. Participants with a contraindication to colonoscopy and polypectomy.
4. Patients with inflammatory bowel disease or gastrointestinal polyposis.
5. Lesions with submucosal invasion and those suspected of being cancerous at the preprocedural diagnostic evaluation.
6. Patients with pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 982 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Complete resection rate | Up to 5-7 days from operation day
  The polyps and the two biopsies from the margin will be sent to the pathologist for further analysis. Two independent experienced pathologists will evaluate the samples separately and both are blinded to the technique performed for polypectomy. Complete resection rate is defined as the negative pathological evaluation of two biopsies obtained from the margin.

SECONDARY OUTCOMES:
Postoperative delayed bleeding rate | Up to 14 days from operation day
  Incidence of bleeding requiring endoscopic hemostasis intervention within 14 days after surgery
Intraoperative bleeding rate | Up to 1 minute from the time the polyp is resected
  Immediate bleeding is defined as bleeding persists >60s after polypectomy according to the ESGE recommendations (2017) and requires for endoscopic intervention.
En bloc resection rate | Up to 7 days when the pathologists finish the evaluations.
  The lesion is removed at one time, and the integrity of the specimen is maintained
Operation time | From the snare/ injection needle exits the working channel to leaving the wound.
  CSP: the time from the time the snare exits the working channel to leaving the wound. Hsp: time from the injection needle leaving the working channel to leaving the wound
Other related postoperative complications | Up to 48 Hours from the time the polyp is resected
  Perforation, infection, electrocoagulation syndrome, etc
Number of metal clips used | The time when the operation is completed
  Whether metal clips are used for hemostasis, and the number of metal clips

CONTACTS AND LOCATIONS:
Overall Officials: Duowu Zou, PHD/MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Gastroenterolog, Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No